CLINICAL TRIAL: NCT03644823
Title: Combinatory ImmunoTherapy-1 (Com-IT-1) Irradiation and PD-1 Blockade in Locally Advanced / Advanced NSCLC
Acronym: COM-IT-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Åslaug Helland, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COM-IT-1
Record Dates: First submitted 2018-02-06; First posted 2018-08-23 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: radiotherapy; PD1-inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PDL1-inhibitor and radiotherapy (Experimental): PDL1-inhibitor (Atezolizumab) and Radiotherapy (6 Gy x 3)
  Interventions: Drug: Atezolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Atezolizumab — PDL1- inhibitor
  Other Names: Tecentriq
Radiation: Radiotherapy — 6 Gy x 3

SUMMARY:
In this study, the investigators will investigate toxicity in patients treated with a Programmed cell death protein 1 (PD-1) inhibitor and radiotherapy. Patients with advanced Non-Small Cell Lung Cancer (NSCLC) can be included when treatment with a PD-1 inhibitor is indicated according to national guidelines. Included patients will receive stereotactic radiotherapy to one or two tumour lesion(s) in addition to the PD-1 inhibitor, and toxicity is the primary endpoint.

DETAILED DESCRIPTION:
This phase II study will investigate NSCLC patients (stage III-IV, palliative treated) where treatment with a PD1-inhibitor is indicated according to national guidelines. Patients will be treated with a check-point inhibitor combined with radiotherapy (6 Gy x 3) towards lesions (1-2). Atezolizumab is available and reimbursed in the public health system. The radiotherapy dosing is significantly lower than standard stereotactic radiotherapy, and is in accordance with other studies reported in ClinicalTrials.gov. Such a fractionation will putatively induce immunogenic cell death, while being a safe treatment, not likely to induce significant side effects.

Whereas the primary endpoint in our clinical study will be toxicity, the secondary endpoints include response rates, overall survival, safety and tolerability, quality of life, progression-free survival and duration of response. In addition, exploratory endpoints will include immunological response, tumor evolution and dynamics in the tumor microenvironment during treatment, imaging, and biomarkers of clinical response.

ELIGIBILITY:
Inclusion Criteria:

5.1.1 Subject Inclusion Criteria

* Age >18 years
* Advanced NSCLC
* Adequate newly obtained core or excisional biopsy of a recurrent tumor lesion
* Adequate is defined as a biopsy with at least 5 sections tumour tissue available.
* Measurable disease according to RECIST criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy > 3 months
* A tumour lesion suitable for radiotherapy treatment
* Adequate organ function based on clinical examination and lab values (Hb >9.0, Leucocytes > 2.0, Trc > 100, AST/ALT <3 ULN)
* Women must not be pregnant or breastfeeding
* WOCBP should use an adequate highly effective method to avoid pregnancy for 23 weeks
* For the purpose of this document, a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

  * Highly effective contraception methods includes methods that can achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include:
  * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  * intrauterine device (IUD)
  * intrauterine hormone-releasing system ( IUS)
  * bilateral tubal occlusion
  * vasectomised partner
* sexual abstinence ___________________________________
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for a period of 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo five half-lives
* Previously untreated or treated NSCLC pts, where treatment with PD1-inhibitor in indicated according to national guidelines.

Exclusion Criteria:

5.1.2 Subject Exclusion Criteria

* Disease suitable for curative salvage surgery
* Treatment with any investigational medicinal product (IMP) that may interfere with the study treatment, within 2 weeks prior to first administration of study drug.
* Significant cardiac, pulmonary or other medical illness that would limit activity or survival
* Pregnancy or lactation.
* Patients with EGFR-mutation or ALK-translocation not treated with tyrosine kinase inhibitor previously
* Known hypersensitivity to any of the components of the investigational product
* Patients who test positive for hepatitis B, C or HIV.
* Known active brain metastases. Patients with stable / treated brain metastases can be included.
* Diagnosis of immunodeficiency or medical condition requiring high doses (>30 mg prednisolone daily) of systemic steroids or other forms of immunosuppressive therapy
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events graded according to NCI CTCAE v4.0 | 24 months
  Adverse events will be graded according to the NCI-CTCAE version 4.0, and registered

SECONDARY OUTCOMES:
Progression free survival | 24 months
  Survival data and responses will be evaluated from tumor assessments per RECIST v1.1, or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Åslaug Helland, Principal Investigator — Radium Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No